CLINICAL TRIAL: NCT07145593
Title: Gamma Transcranial Alternating Current Stimulation in Attention Deficit Hyperactivity Disorder
Brief Title: Gamma tACS in Attention-Deficit/Hyperactivity Disorder
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, FATMA AYDIN, Principal Investigator, Medipol University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: E-10840098-202.3.02-4603
Record Dates: First submitted 2025-07-30; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: gamma; EEG; tACS
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 80 Hz Group (Experimental): Transcranial alternating current stimulation (tACS) at 80 Hz gamma frequency will be applied to the bilateral dorsolateral prefrontal cortex (DLPFC). Each session will last 20 minutes. A total of five sessions will be conducted.
  Interventions: Device: Application tACS- 80 Hz
- 6-80 Hz Group (Experimental): Transcranial alternating current stimulation (tACS) at 6-80 Hz theta- gamma frequency will be applied to the bilateral dorsolateral prefrontal cortex (DLPFC). Each session will last 20 minutes. A total of five sessions will be conducted.
  Interventions: Device: Application TACS - (6-80 Hz)
- Sham Group (Sham Comparator): Transcranial alternating current stimulation (tACS) sham will be applied to the the bilateral dorsolateral prefrontal cortex (DLPFC). Each session will last 20 minutes. A total of five sessions will be conducted.
  Interventions: Device: Application TACS- Sham
- 40 Hz Group (Experimental): Transcranial alternating current stimulation (tACS) at 40 Hz gamma frequency will be applied to the bilateral dorsolateral prefrontal cortex (DLPFC). Each session will last 20 minutes. A total of five sessions will be conducted.
  Interventions: Device: Application tACS -40 Hz
- Individual Gamma Group (Experimental): Transcranial alternating current stimulation (tACS) at ındividual gamma frequency will be applied to the bilateral dorsolateral prefrontal cortex (DLPFC). Each session will last 20 minutes. A total of five sessions will be conducted.
  Interventions: Device: Application TACS- Individual Gamma Hz

INTERVENTIONS:
Device: Application tACS- 80 Hz — In this study, a single 20-minute session of tACS will be administered over the bilateral dorsolateral prefrontal cortex (DLPFC) at various gamma frequencies (80 Hz).The anodal surface electrode will be placed over the left DLPFC (F3 according to the 10-20 system), and the cathodal electrode over the right DLPFC (F4).
  Arms: 80 Hz Group
Device: Application tACS -40 Hz — In this study, a single 20-minute session of tACS will be administered over the bilateral dorsolateral prefrontal cortex (DLPFC) at gamma frequencies (40 Hz). The anodal surface electrode will be placed over the left DLPFC (F3 according to the 10-20 system), and the cathodal electrode over the right DLPFC (F4).
  Arms: 40 Hz Group
Device: Application TACS - (6-80 Hz) — In this study, a single 20-minute session of tACS will be administered over the bilateral dorsolateral prefrontal cortex (DLPFC) at theta- gamma coupling frequencies ( 6-80 Hz). The anodal surface electrode will be placed over the left DLPFC (F3 according to the 10-20 system), and the cathodal electrode over the right DLPFC (F4).
  Arms: 6-80 Hz Group
Device: Application TACS- Individual Gamma Hz — In this study, a single 20-minute session of tACS will be administered over the bilateral dorsolateral prefrontal cortex (DLPFC) at individual gamma frequencies . The anodal surface electrode will be placed over the left DLPFC (F3 according to the 10-20 system), and the cathodal electrode over the right DLPFC (F4).
  Arms: Individual Gamma Group
Device: Application TACS- Sham — In this study, a single 20-min tACS session will be applied over the bilateral dorsolateral prefrontal cortex (DLPFC) in a sham application. The anodal surface electrode will be placed over the left DLPFC (F3 of the 10-20 system) and the cathodal electrode will be placed over the right DLPFC (F4).
  Arms: Sham Group

SUMMARY:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a common neurodevelopmental disorder characterized by symptoms of inattention, impulsivity, and hyperactivity. These symptoms are often associated with impairments in executive functions and working memory, which are essential for goal-directed behavior and cognitive control. Deficits in these domains can significantly hinder individuals' academic, social, and daily functioning. Gamma oscillations (30-80 Hz) play a crucial role in cognitive integration, attention, and memory processes, and are thought to emerge from the balance between excitatory and inhibitory neuronal activity.

Transcranial Alternating Current Stimulation (tACS) is a non-invasive brain stimulation technique that modulates neuronal activity through rhythmic electrical currents. Recent studies suggest that gamma-frequency tACS applied to the prefrontal cortex can enhance cognitive performance and attentional processes. In individuals with ADHD, disrupted gamma connectivity and reduced regional gamma power have been associated with attentional deficits. Therefore, gamma tACS may modulate both regional activity and long-range functional connectivity, offering a promising neuromodulation strategy to alleviate ADHD symptoms.

In this context, the present study aims to investigate the effects of bilateral gamma-frequency tACS applied to the prefrontal cortex on attention and executive function performance in individuals with ADHD. Changes in gamma oscillatory activity will be measured using EEG to assess the neurophysiological impacts of stimulation. The study seeks to evaluate whether gamma tACS can serve as a targeted, evidence-based intervention to address the neurofunctional deficits observed in ADHD, potentially offering a novel therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 40 years of age
* Receiving an ADHD diagnosis
* Scoring above 25 on the Montreal Cognitive Assessment (MoCA)
* Being right-handed

Exclusion Criteria:

* Use of medications with sedative or stimulant effects
* Presence of metal brain implants or a pacemaker

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Öktem Verbal Memory Test | Pre-tACS Baseline (prior to stimulation) / Post-tACS (within 30 minutes after stimulation)
  Öktem Verbal Memory Test is a test of verbal memory processes, developed and validated by Öktem in 1992. It is designed to measure various variables related to memory.
Forward and Backward Digit Span | Pre-tACS Baseline (prior to stimulation) / Post-tACS (within 30 minutes after stimulation)
  This test, which is a subtest of the Wechsler Memory Scale, was developed to assess overall attention. It consists of two stages. The first stage evaluates the forward digit span, composed of random sequences ranging from 2 to 8 digits. In the second stage, the backward digit span is assessed using random sequences of 2 to 7 digits. In the first stage, numbers are read aloud with one-second intervals, and participants are expected to repeat the sequences exactly as presented. In the second stage, numbers are again read with one-second intervals, but participants are required to repeat the digits in reverse order. The test is terminated if the participant makes consecutive errors. The forward digit span assesses sustained attention, while the backward span also evaluates working memory performance.
Verbal fluency tests | Pre-tACS Baseline (prior to stimulation) / Post-tACS (within 30 minutes after stimulation)
  Verbal fluency tests measure the ability to generate words within a specific category over a limited time period. Verbal fluency performance has been associated not only with general language skills and semantic memory functions but also with executive functions such as attention, working memory, and processing speed. In this study, semantic and phonemic fluency tasks will be used.
Resting State EEG and TASK EEG | Pre-tACS Baseline (prior to stimulation) / Post-tACS (within 30 minutes after stimulation)
  The EEG recordings of the participants will be conducted using a BrainAmp 64-channel DC system. A 64-channel EasyCap will be used. AFz will serve as the ground electrode, and FCz will be used as the reference electrode. Impedance values will be maintained below 10 kOhm. EEG data will be recorded using the BrainVision Recorder software (Brain Products, Munich, Germany) with a band-pass filter set between 0.01 and 250 Hz.A 4-minute eyes-open and a 4-minute eyes-closed resting-state EEG recording will be conducted. EEG will also be recorded during the 2-back task and the memory task. 2-back Task: A visual n-back task will be administered to assess working memory. The task load will consist of 8-minute sessions. Memory Task: The memory task, which involves both encoding and retrieval of episodic information, will be examined using a visual memory paradigm presented to the participants.

OTHER OUTCOMES:
The Self-Reported Attention Deficit Scale | Baseline
  The Self-Reported Attention Deficit Scale is one of the screening tools developed by the World Health Organization (WHO) to identify mental disorders. The scale consists of two subscales: "attention deficit" and "hyperactivity/impulsivity," each comprising nine items. These questions are designed to assess how frequently each symptom has occurred over the past six months. Responses are scored on a scale ranging from 0 to 4, where 0 indicates "never," 1 indicates "rarely," 2 indicates "sometimes," 3 indicates "often," and 4 indicates "very often."
Montreal Cognitive Assessment (MoCA) | Baseline
  MoCA is a widely used tool designed to evaluate individuals' cognitive functions. The test scores range from a minimum of 0 to a maximum of 30. In the MoCA, higher scores indicate better cognitive performance, while lower scores may suggest the presence of cognitive impairment. In clinical practice, a score of 26 or above is generally considered indicative of normal cognitive functioning, whereas scores below 26 may reflect mild cognitive impairment. Additionally, it is recommended to add 1 point to the total score for individuals with 12 years of education or less. Scores between 18-25 are typically associated with mild cognitive impairment, scores between 10-17 with moderate impairment, and scores between 0-9 with severe cognitive impairment. However, MoCA test results should always be interpreted in conjunction with comprehensive clinical evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfü Hanoğlu, Study Director — Medipol University; Suat Yılmaz, Principal Investigator — Medipol University; Gülsüm Uzer, Principal Investigator — Medipol University
Locations (1):
- Medipol University Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided